CLINICAL TRIAL: NCT02023242
Title: A Prospective, Multicenter, Randomized Comparison of the Hydrus to the iStent® for Lowering Intraocular Pressure in Primary Open Angle Glaucoma
Brief Title: Comparing Effectiveness of the Hydrus Microstent (TM) to Two iStents to Lower IOP in Phakic Eyes
Acronym: COMPARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ivantis, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CP-12-001
Record Dates: First submitted 2013-12-23; First posted 2013-12-30 (Estimated); Results first posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Primary Open Angle Glaucoma; Pseudoexfoliative Glaucoma; Pigmentary Glaucoma
Keywords: Primary open angle glaucoma; POAG; Pseudoexfoliative glaucoma; PXG; Pigmentary glaucoma; PG; Hydrus
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydrus Microstent (Experimental): Patients randomized to the Hydrus Microstent .
  Interventions: Device: Hydrus Microstent
- iStent Trabecular Micro Bypass (Active Comparator): Patients randomized to the iStent Trabecular Micro Bypass
  Interventions: Device: iStent Trabecular Micro Bypass

INTERVENTIONS:
Device: Hydrus Microstent — Device inserted into Schlemm's canal to enhance aqueous flow from the anterior chamber.
  Arms: Hydrus Microstent
Device: iStent Trabecular Micro Bypass — Device inserted into Schlemm's canal to enhance aqueous flow from the anterior chamber.
  Arms: iStent Trabecular Micro Bypass

SUMMARY:
This clinical trial compares two implantable devices intended to lower the pressure inside the eye of glaucoma patients.

DETAILED DESCRIPTION:
This is a prospective, multicenter, single-masked, randomized clinical trial comparing the Hydrus Microstent to two iStent implants for the reduction of intraocular pressure in phakic patients with a positive diagnosis of primary open angle glaucoma, pseudoexfoliative glaucoma, or pigmentary dispersion glaucoma. Post-operative follow-up visits will be conducted at regular intervals.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of primary open angle glaucoma (POAG), Pseudoexfoliative (PXG) glaucoma, or Pigmentary glaucoma (PG)
* A phakic lens with BCVA of 20/30 or better

Exclusion Criteria:

* Forms of primary or secondary glaucoma not listed above
* Prior glaucoma surgery in the study eye

Ages: 45 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2012-10; Primary Completion 2017-08 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julian Garcia Feijoo, Prof. Med., Principal Investigator — Madrid, Spain
Locations (1):
- Contact Richard Hope at Ivantis, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened and enrolled at 12 investigational sites located outside of the United States
Pre-assignment Details: 152 patients were randomized
Groups:
- Hydrus Microstent: Subjects underwent 1 Hydrus implantation
- iStent Trabecular Micro Bypass: Subjects underwent 2 iStents implantation
Period: Overall Study
Arm/Group | Hydrus Microstent | iStent Trabecular Micro Bypass
Started | 75 | 77
Completed | 72 | 75
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) - All participants randomized and grouped according to their randomization assignment
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrus Microstent | iStent Trabecular Micro Bypass | Total
Number analyzed (Participants) | 75 | 77 | 152
Age, Continuous [Median (Standard Deviation); unit: years] | 67.5 (10.3) | 66.5 (9.5) | 67.0 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 45 | 86
  Male | 34 | 32 | 66
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian/White European | 49 | 49 | 98
  Black or African Descent | 1 | 3 | 4
  Asian | 11 | 11 | 22
  Native North American | 0 | 0 | 0
  Hispanic/Latino/Central & So American Origin | 14 | 13 | 27
  Other | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Unmedicated IOP </= 19 mmHg at 12 Months
Description: Percentage of subjects with IOP </= 19 mmHg and without the use of ocular hypotensive medications at 12 months
Time Frame: 12 months
Population: Intent-to-Treat (ITT)
Measure: Number; unit: percentage of participants
Arm/Group | Hydrus Microstent | iStent Trabecular Micro Bypass
Number analyzed (Participants) | 73 | 75
percentage of participants | 34.2 | 13.3

2. Secondary Outcome: The Percentage of Subjects Who Are Not Using Ocular Hypotensive Medications at 12 and 24 Months
Description: The percentage of subjects who are not using ocular hypotensive medications at 12 and 24 months
Time Frame: 12 & 24 Months
Population: Intent-to-Treat (ITT). Number of Participants Analyzed at 24 Months in the Hydrus Microstent arm are different than at 12 Months due to patients lost to follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Hydrus Microstent | iStent Trabecular Micro Bypass
Number analyzed (Participants) | 73 | 75
percentage of participants
  12 Months | 46.6 | 24.0
  24 Months: number analyzed (Participants) | 71 | 75
  24 Months | 38.0 | 18.7

3. Secondary Outcome: Mean Medication Use at 12 and 24 Months
Description: The mean medication use at 12 and 24 months
Time Frame: 12 & 24 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: number of medications
Arm/Group | Hydrus Microstent | iStent Trabecular Micro Bypass
Number analyzed (Participants) | 73 | 75
number of medications
  12 Months | 0.99 (1.07) | 1.69 (1.37)
  24 Months: number analyzed (Participants) | 71 | 75
  24 Months | 1.23 (1.15) | 1.91 (1.36)

4. Secondary Outcome: Unmedicated IOP </= 19 mmHg at 24 Months
Description: Percentage of subjects with IOP </= 19 mmHg and without the use of ocular hypotensive medications at 24 months
Time Frame: 24 Months
Population: Intent-to-Treat (ITT). Number of Participants Analyzed at 24Months in the Hydrus Microstent arm are different than at 12 Months due to patients lost to follow-up
Measure: Number; unit: percentage of participants
Arm/Group | Hydrus Microstent | iStent Trabecular Micro Bypass
Number analyzed (Participants) | 71 | 75
percentage of participants | 23.9 | 13.3

5. Secondary Outcome: Unmedicated IOP </= 18 mmHg at 12 Months
Description: Percentage of subjects with IOP </= 18 mmHg and without the use of ocular hypotensive medications at 12 months
Time Frame: 12 months
Population: Intent-to-Treat (ITT)
Measure: Number; unit: percentage of participants
Arm/Group | Hydrus Microstent | iStent Trabecular Micro Bypass
Number analyzed (Participants) | 73 | 75
percentage of participants | 30.1 | 9.3

ADVERSE EVENTS:
Time Frame: 24 Months
Description: An adverse event is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, users or other persons, whether or not related to the investigational medical device. All subjects who have been exposed to the study treatment were evaluated for adverse events.
Arm/Group | Hydrus Microstent | iStent Trabecular Micro Bypass
All-Cause Mortality (participants affected / at risk) | 0/75 | 1/77
Serious Adverse Events (participants affected / at risk) | 7/75 | 14/77
Other Adverse Events (participants affected / at risk) | 24/75 | 23/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrus Microstent (N=75) | iStent Trabecular Micro Bypass (N=77)
BCVA loss >/= 2 lines ETDRS >/= 3 months (Eye disorders) | 0 (0) | 2 (2)
Cataract (Eye disorders) | 3 (3) | 2 (2)
IOP Increase (Eye disorders) | 0 (0) | 1 (1)
IOP increase (>=10 mmHg than BL >= 1M) (Eye disorders) | 0 (0) | 1 (1)
Inflammation lasting >1M (Eye disorders) | 0 (0) | 1 (1)
Proliferative Diabetic Retinopathy (Eye disorders) | 1 (1) | 0 (0)
Uncontrolled Glaucoma (Eye disorders) | 0 (0) | 7 (8)
Wet Age Related Macular Degeneration (Eye disorders) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrus Microstent (N=75) | iStent Trabecular Micro Bypass (N=77)
BCVA loss >= 2 lines ETDRS >= 3M (Post-Operative) (Eye disorders) | 5 (5) | 9 (9)
Device Obstruction (Post-Operative) (Eye disorders) | 6 (6) | 10 (10)
PAS with Device Obstruction (Post-Operative) (Eye disorders) | 5 (5) | 1 (1)
PAS without Device Obstruction (Post-Operative) (Eye disorders) | 8 (8) | 3 (3)
Device Malposition (Intraoperative) (Eye disorders) | 2 (2) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"If the Clinical Investigation is multi-centered, any publication based on the results obtained at the Investigation Site (or a group of sites) shall not be made before the first multi-center publication."

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-03-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT02023242/Prot_SAP_000.pdf